CLINICAL TRIAL: NCT05274074
Title: Improving Care Partner Outcomes Through Positive Connections
Brief Title: Social-LEAF Life Enhancing Activities for Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Benzi Kluger, MD, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 375254; P30AG064103 (NIH)
Record Dates: First submitted 2022-01-27; First posted 2022-03-10 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Social Connectedness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait-List Control (No Intervention): The wait-list control had a 6 week waiting period after which they received the Social LEAF intervention
- Intervention (Experimental): Social LEAF is an adaptation of the Life Enhancing Activities for Family Caregivers program to focus on social relationships and loneliness.We utilized the Life Enhancing Activities or Caregivers (LEAF) intervention to display that social networks' can be used as a means of reinforcing the positive life skills of the intervention; and that these same skills will enhance social networks, increase mutual satisfaction in social interactions, and boost motivation to reach out to others, thus combatting social isolation.
  This group received the intervention for 6 weeks and we looked at maintenance 6 weeks after the end of the intervention.
  Interventions: Behavioral: Social LEAF

INTERVENTIONS:
Behavioral: Social LEAF — Social LEAF is an adaptation of the Life Enhancing Activities for Family Caregivers program to focus on social relationships and loneliness. Social LEAF is a six-session group program provided by video-conference that teaches caregivers coping skills to improve social relationships and social connection. Social LEAF is delivered in groups of up to 10 caregivers via videoconference and will consist of six weekly hour-long discussion-based classes to teach positive coping skills around improving social relationships. Each week will focus on a skill from the original LEAF study adapted to the group and social context.
  Arms: Intervention

SUMMARY:
This study examines a behavioral intervention to improve social connection and reduce loneliness for caregivers of a loved one with Dementia with Lewy Bodies (DLB).

DETAILED DESCRIPTION:
The objective of the Social-LEAF study is to examine psychological mechanisms whereby Social LEAF delivered in a group and via video call reduces loneliness and improves positive emotions for older caregivers of loved ones with DLB. This is an 18-month Stage 2 study examining Social LEAF, which is strengths-based and teaches positive coping skills focused on improving social relationships and is delivered remotely in a group format. These two adaptations to the original LEAF intervention are included to provide a more potent means of improving social connection. A pilot phase with up to 20 caregivers (Aim 1) will address these adaptations regarding feasibility, acceptability, and signal for reducing loneliness, with refinements as needed. A second phase (Aims 2 and 3) will involve a randomized trial comparing Social LEAF to control (30 caregivers in each arm) on loneliness (primary outcome), positive affect (mechanism), and social engagement (mechanism). Data will also be collected on acceptability and perceived benefits using mixed methods.

Aim 1 is to refine the LEAF intervention to target social relationships and loneliness.

Aim 2 is to examine feasibility and acceptability of Social LEAF for DLB caregivers.

Aim 3 is to examine efficacy of Social LEAF in reducing loneliness, increasing positive affect, and increasing social engagement.

ELIGIBILITY:
Inclusion criteria:

* Must be a primary care partner of a person that has been clinically diagnosed with Dementia with Lewy Bodies (DLB) or Parkinson's Disease Dementia, and has access to high-speed internet connection at home or in a location where they can speak privately with a facilitator. iPads and a hotspot will be given to those who lack internet and a sufficient mobile device but show willingness to participate. The iPads and hotspot will be returned to the study team once study procedures have concluded. Must be willing and ready to begin the intervention either immediately or in 6 weeks depending on which group they are randomly selected to be in.
* Must begin LEAF procedures as soon as consented to the study. Has not taken part in Aim 1 of the study.
* Will have waited the 6-week period before starting LEAF procedures after consenting and has not taken part in Aim 1 of the study.

Exclusion Criteria:

* Not a primary care partner of a person with DLB. Is a primary care partner of someone who has not been clinically diagnosed with DLB. Cannot speak English or provide clear and concise consent to the project.
* Has not started LEAF procedures at the beginning and has taken part in Aim 1 of the study.
* Has started/taken part in the LEAF procedures at the beginning and also has taken part in Aim 1 of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-07-23 (Actual); Study Completion 2023-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data will be made available upon request and after review by the study team.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of main manuscript
Access Criteria: Requesting investigators will need to provide a rationale for their request and plan for results. Depending on request, a Data User Agreement may also be required.

RESULTS

PARTICIPANT FLOW:
Groups:
- Wait-List Control: The wait-list control had a 6 week waiting period after which they had the option of doing the intervention.
- Intervention: We will be utilizing the Life Enhancing Activities or Caregivers (LEAF) intervention to display that social networks' can be used as a means of reinforcing the positive life skills of the intervention; and that these same skills will enhance social networks, increase mutual satisfaction in social interactions, and boost motivation to reach out to others, thus combatting social isolation.
  This group received the intervention for 6 weeks and we looked at maintenance 6 weeks after the end of the intervention.
  Social LEAF: Social LEAF is an adaptation of the Life Enhancing Activities for Family Caregivers program to focus on social relationships and loneliness. Social LEAF is a six-session group program provided by video-conference that teaches caregivers coping skills to improve social relationships and social connection. Social LEAF is delivered in groups of up to 10 caregivers via videoconference and will consist of six weekly hour-long discussion-based classes to teach positive coping skills around improving social relationships. Each week will focus on a skill from the original LEAF study adapted to the group and social context.
Period: Overall Study
Arm/Group | Wait-List Control | Intervention
Started | 29 | 29
Completed | 26 | 24
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wait-List Control | Intervention | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (12) | 67 (13) | 67 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 28 | 26 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 26 | 27 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58
PROMIS Positive Affect [Mean (Standard Deviation); unit: units on scale] — The Patient Reported Outcomes Measurement Information System (PROMIS)- Positive Affect is a 15-item scale measuring momentary positive affective experiences over the past 7 days. It is a five-point Likert-type scale (i.e.,"not at all, a little bit, somewhat, quite a bit, very much"). Scores are summed to create a raw score. Individual items are positively skewed with 5 options from "Not at all" to "Very much." Higher scores indicate better positive affect and are a better outcome. Population: 3 participants did not complete the baseline Positive Affect Measure
  units on scale
    number analyzed (Participants) | 27 | 28 | 55
    (all) | 41.9 (8.8) | 45.5 (8.5) | 43.7 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Outcome Measurement Information System (PROMIS )Positive Affect
Description: Change in the Patient Reported Outcomes Measurement Information System (PROMIS)- Positive Affect from Baseline to Week 6. This is a 15-item scale measuring momentary positive affective experiences over the past 7 days. It is a five-point Likert-type scale (i.e.,"not at all, a little bit, somewhat, quite a bit, very much") resulting in 15-75 scale. Scores are summed to create a raw score. Individual items are positively skewed with 5 options from "Not at all" to "Very much." Higher scores indicate better positive affect and are a better outcome.
Time Frame: Week 6
Population: Caregivers of persons with Lewy-body dementia were randomized to intervention and wait-list control groups. Nine participants did not complete either baseline or the 6-week measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Intervention: We utilized the Life Enhancing Activities or Caregivers (LEAF) intervention to display that social networks' can be used as a means of reinforcing the positive life skills of the intervention; and that these same skills will enhance social networks, increase mutual satisfaction in social interactions, and boost motivation to reach out to others, thus combatting social isolation.
  This group received the intervention for 6 weeks and we looked at outcomes at week 6 post-intervention.
  Social LEAF: Social LEAF is an adaptation of the Life Enhancing Activities for Family Caregivers program to focus on social relationships and loneliness. Social LEAF was a six-session group program provided by video-conference that taught caregivers coping skills to improve social relationships and social connection. Social LEAF was delivered in groups of up to 10 caregivers via videoconference and consisted of six weekly hour-long discussion-based classes to teach positive coping skills around improving social relationships. Each week focused on a skill from the original LEAF study adapted to the group and social context.
Arm/Group | Wait-List Control | Intervention
Number analyzed (Participants) | 25 | 24
units on a scale | -1.7 [-5.1 to 1.7] | -0.3 [-3.8 to 3.1]
Statistical Analysis 1: Comparison: Wait-List Control vs Intervention; Test type: Superiority; p = 0.57, Regression, Linear; Mean Difference (Net) = 1.4, 95% CI 2-sided [-3.4 to 6.2]

2. Secondary Outcome: Berkman-Syme Social Network Index
Description: Change in the Berkman-Syme Social Network Index from baseline to week 6. This scale is used to measure social isolation and loneliness and includes subjective experiences of connection to contacts. This measure is a questionnaire to assess the type, size, closeness, and frequency of contacts in a respondent's current social network. This index is the sum of four binary items (Married (no = 0; yes = 1); close friends and relatives (0-2 friends and 0-2 relatives = 0; all other scores = 1); group participation (no = 0; yes = 1); participation in religious meetings or services (less than or equal to every few months = 0; greater than or equal to once or twice a month = 1)). The total index range is 0-4 with a higher score indicative of better social network.
Time Frame: Week 6
Population: Caregivers of persons with Lewy-body dementia were randomized to intervention and wait-list control groups. Eight participants did not complete either baseline or the 6-week measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Intervention: We utilized the Life Enhancing Activities or Caregivers (LEAF) intervention to display that social networks' can be used as a means of reinforcing the positive life skills of the intervention; and that these same skills will enhance social networks, increase mutual satisfaction in social interactions, and boost motivation to reach out to others, thus combatting social isolation.
  This group received the intervention for 6 weeks and we looked at maintenance 6 weeks after the end of the intervention.
  Social LEAF: Social LEAF is an adaptation of the Life Enhancing Activities for Family Caregivers program to focus on social relationships and loneliness. Social LEAF was a six-session group program provided by video-conference that taught caregivers coping skills to improve social relationships and social connection. Social LEAF was delivered in groups of up to 10 caregivers via videoconference and consisted of six weekly hour-long discussion-based classes to teach positive coping skills around improving social relationships. Each week focused on a skill from the original LEAF study adapted to the group and social context.
Arm/Group | Wait-List Control | Intervention
Number analyzed (Participants) | 26 | 24
units on a scale | -0.8 [-1.0 to -0.6] | -0.9 [-1.2 to -0.7]
Statistical Analysis 1: Comparison: Wait-List Control vs Intervention; Test type: Superiority; p = 0.53, Regression, Linear; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.5 to 0.2]

3. Secondary Outcome: Patient Reported Outcome Measurement Information System (PROMIS) Social Isolation
Description: Change in the Patient Reported Outcome Measurement Information System (PROMIS)- Social Isolation from baseline to week 6. This scale assesses perceptions of being avoided, excluded, detached, disconnected from by others. The measure has a Likert Scale (1-5 with 1 being Never and 5 being Always). Raw scores were converted to a T-score, a standardized score with a mean of 50 and a standard deviation of 10. Lower scores indicate lesser social isolation and are therefore a better outcome.
Time Frame: Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Waitlist Control: The wait-list control had a 6 week waiting period after which they had the option of doing the intervention
- Intervention Group: We utilized the Life Enhancing Activities or Caregivers (LEAF) intervention to display that social networks' can be used as a means of reinforcing the positive life skills of the intervention; and that these same skills will enhance social networks, increase mutual satisfaction in social interactions, and boost motivation to reach out to others, thus combatting social isolation.
  This group received the intervention for 6 weeks and we looked at outcomes at week 6 post-intervention.
  Social LEAF: Social LEAF is an adaptation of the Life Enhancing Activities for Family Caregivers program to focus on social relationships and loneliness. Social LEAF was a six-session group program provided by video-conference that taught caregivers coping skills to improve social relationships and social connection. Social LEAF was delivered in groups of up to 10 caregivers via videoconference and consisted of six weekly hour-long discussion-based classes to teach positive coping skills around improving social relationships. Each week focused on a skill from the original LEAF study adapted to the group and social context.
Arm/Group | Waitlist Control | Intervention Group
Number analyzed (Participants) | 26 | 24
units on a scale | 0.9 [-0.7 to 2.5] | -0.1 [-1.7 to 1.6]
Statistical Analysis 1: Comparison: Waitlist Control vs Intervention Group; Test type: Superiority; p = 0.41, Regression, Linear; Mean Difference (Net) = -1.0, 95% CI 2-sided [-3.3 to 1.4]

4. Secondary Outcome: Patient Reported Outcome Measurement Information System (PROMIS) Satisfaction Role Activities
Description: Change in the PROMIS V 2.0 Satisfaction Role Activities from baseline to week 6. This scale assessed caregivers satisfaction level in their participation in relaxation and leisure activities.The measure has a Likert Scale (1-5 with 1 being Not at all and 5 being Very much). Raw scores were converted to a T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher satisfaction and are therefore a better outcome.
Time Frame: Week 6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Intervention Group: We utilized the Life Enhancing Activities or Caregivers (LEAF) intervention to display that social networks' can be used as a means of reinforcing the positive life skills of the intervention; and that these same skills will enhance social networks, increase mutual satisfaction in social interactions, and boost motivation to reach out to others, thus combatting social isolation.
  This group received the intervention for 6 weeks and we looked at maintenance 6 weeks after the end of the intervention.
  Social LEAF: Social LEAF is an adaptation of the Life Enhancing Activities for Family Caregivers program to focus on social relationships and loneliness. Social LEAF was a six-session group program provided by video-conference that taught caregivers coping skills to improve social relationships and social connection. Social LEAF was delivered in groups of up to 10 caregivers via videoconference and consisted of six weekly hour-long discussion-based classes to teach positive coping skills around improving social relationships. Each week focused on a skill from the original LEAF study adapted to the group and social context.
Arm/Group | Waitlist Control | Intervention Group
Number analyzed (Participants) | 26 | 24
units on a scale | -0.1 [-1.8 to 1.6] | -1.0 [-2.9 to 0.8]
Statistical Analysis 1: Comparison: Waitlist Control vs Intervention Group; Test type: Superiority; p = 0.45, Regression, Linear; Mean Difference (Net) = -0.9, 95% CI 2-sided [-3.5 to 1.6]

5. Secondary Outcome: Positive Aspects of Caregiving Scale
Description: Change in the Positive Aspects of Caregiving Scale from baseline to week 6. This scale consists of nine items assessing positive consequences of caregiving, each rated on a 0-4 Likert scale (range of scores 0-36), where a higher score reflects a more positive perception of the caregiving experience.
Time Frame: Week 6
Population: Caregivers of persons with Lewy-body dementia were randomized to intervention and wait-list control groups. Eight participants did not complete either baseline or the 6-week measure.
  Caregivers of persons with Lewy-body dementia were randomized to intervention and wait-list control groups. Eight participants did not complete either baseline or the 6-week measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Wait-List Control | Intervention
Number analyzed (Participants) | 26 | 24
units on a scale | -0.8 [-2.8 to 1.1] | 2.5 [0.4 to 4.6]
Statistical Analysis 1: Comparison: Wait-List Control vs Intervention; Test type: Superiority; p = 0.02, Regression, Linear; Mean Difference (Net) = 3.3, 95% CI 2-sided [0.5 to 6.2]

6. Secondary Outcome: University of California Los Angeles (UCLA) Loneliness Scale
Description: Change in the UCLA Loneliness scale from baseline to week 6. This scale produces a continuous score of the degree to which participants endorse loneliness. The measure has 20 items with a Likert scale of 1-4 with 1 being Never and 4 being Always resulting in a 20-80 scale. Lower scores indicate better outcome.
Time Frame: Week 6
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Wait-List Control | Intervention
Number analyzed (Participants) | 26 | 24
units on a scale | 0.6 [-2.2 to 3.5] | -0.2 [-3.1 to 2.8]
Statistical Analysis 1: Comparison: Wait-List Control vs Intervention; Test type: Superiority; p = 0.69, Regression, Linear; Mean Difference (Net) = -0.8, 95% CI 2-sided [-4.9 to 3.3]

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Wait-List Control: The wait-list control had a 6 week waiting period after which they received the intervention.
- Intervention: We utilized the Life Enhancing Activities or Caregivers (LEAF) intervention to display that social networks' can be used as a means of reinforcing the positive life skills of the intervention; and that these same skills will enhance social networks, increase mutual satisfaction in social interactions, and boost motivation to reach out to others, thus combatting social isolation.
  This group received the intervention for 6 weeks and we looked at outcomes at week 6 post-intervention.
Arm/Group | Wait-List Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

LIMITATIONS AND CAVEATS:
This is a small pilot trial. The intent was primarily to assess feasibility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT05274074/Prot_002.pdf
  • Statistical Analysis Plan (2025-01-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT05274074/SAP_003.pdf
  • Informed Consent Form (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT05274074/ICF_004.pdf